CLINICAL TRIAL: NCT04675489
Title: Patient Satisfaction and Visual Outcomes After Bilateral Implantation of a Novel Non-Diffractive Extended Vision Toric Intraocular Lens
Brief Title: Visual Outcomes After Vivity Toric IOL Implantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting
Sponsor: EVP Eye Care (Other)
Collaborators: Alcon Research (Industry); Icon Eye Care (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-01
Record Dates: First submitted 2020-11-13; First posted 2020-12-19 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2020-12

CONDITIONS: Refractive Assessment
Keywords: Vivity; Extended Vision Toric Intraocular Lens; Patient satisfaction and visual outcomes
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Subjects to receive bilateral implantation of Vivity Extended Vision Toric Intraocular Lens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vivity Toric IOL (Other): Patients with cataract that had phacoemulsification and Vivity Toric IOL implantation.
  Interventions: Other: Procedure: Vivity Toric IOL

INTERVENTIONS:
Other: Procedure: Vivity Toric IOL — The U.S. Food and Drug Administration (FDA) has granted approval of Alcon's Vivity Toric Extended Vision intraocular lens (IOL) for cataract patients. This innovative lens is an extended depth of focus IOL that has been reported to result in fewer visual disturbances than diffractive IOLs.

SUMMARY:
The purpose of this study is to evaluate patient satisfaction after bilateral implantation of Vivity Toric Extended Vision Intraocular lens and visual outcomes.

DETAILED DESCRIPTION:
To evaluate and report outcomes including postoperative uncorrected visual acuity, postoperative best corrected visual acuity, postoperative refractive error, and IOL rotational stability after Vivity Toric Extended Vision intraocular lens (IOL) implantation.

ELIGIBILITY:
Inclusion Criteria:

* Calculated lens power within study IOL range of 15.0 diopters to 25.0 diopters and toric range of T3 to T6
* Willing and able to comprehend informed consent form and to complete 1 day and 3-4 month postoperative visit
* Potential postoperative best corrected distance visual acuity of 20/20 or better in each eye based on medical opinion of investigator

Exclusion Criteria:

* Ocular pathology or comorbidity that could reduce potential postoperative best corrected distance visual acuity
* Ocular trauma or zonular weakness/instability
* Diagnosis of glaucoma or high-risk glaucoma suspect
* Previous refractive surgery
* Unreliable preoperative biometry measurements
* Severe dry eye or ocular surface disease

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Monocular visual acuity at distance | 4 months
  Monocular uncorrected distance visual acuity
Binocular visual acuity at distance | 4 months
  Binocular uncorrected distance visual acuity
Monocular best corrected distance visual acuity | 4 months
  Monocular best corrected distance visual acuity
Binocular best corrected distance visual acuity | 4 months
  Binocular best corrected distance visual acuity
Monocular best distance-corrected intermediate visual acuity | 4 months
  Monocular best distance-corrected intermediate visual acuity
Binocular best distance-corrected intermediate visual acuity | 4 months
  Binocular best distance-corrected intermediate visual acuity
Monocular best distance-corrected near visual acuity | 4 months
  Monocular best distance-corrected near visual acuity
Binocular best distance-corrected near visual acuity | 4 months
  Binocular best distance-corrected near visual acuity

SECONDARY OUTCOMES:
Residual refractive cylinder | 4 months
  Manifest postoperative refractive cylinder (measured in diopters, with a phoropter) after cataract surgery and IOL implantation.

CONTACTS AND LOCATIONS:
Overall Officials: James Fox, MD, Principal Investigator — Icon Eye Care
Locations (1):
- Icon Eye Care, Grand Junction, Colorado, United States

IPD SHARING:
Plan to Share IPD: No